CLINICAL TRIAL: NCT01991171
Title: Effectiveness of the Kinesio Taping® in Activation of Quadriceps Muscle and Reflex Inhibition of Hamstrings Muscle: Randomized Controlled Trial
Brief Title: Effectiveness of the Kinesio Taping® in Muscle Activation
Acronym: EKTAQRIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Mauricio Antonio da Luz Junior, Effectiveness of the Kinesio Taping® in Activation of Quadriceps Muscle and Reflex Inhibition of Hamstrings Muscle: Randomized Controlled Trial., Paulista University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE14385813.1.0000.5512; 250.259 (Other: Paulista University)
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Muscle Atrophy
Keywords: kinesio taping; Muscle activation; Muscle inhibition
MeSH Terms: conditions — Muscular Atrophy | interventions — Bandages; Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kinesio Taping (Experimental): Participant will receive application of Kinesiotaping in their thigh on quadriceps muscle
  Interventions: Other: Kinesio Taping
- Kinesio Taping Placebo (Placebo Comparator): Participant will receive application of placebo Kinesiotaping in their thigh on quadriceps muscle
  Interventions: Other: Kinesio Taping
- Control Group (No Intervention): This participants will not receive intervention

INTERVENTIONS:
Other: Kinesio Taping — Kinesiotaping intervention is based upon the use of specific elastic tapes (known as Kinesio Tex Gold) that are applied with a certain amount of tension fixed to the skin of patients with the target muscles in a stretched position. The tapes will be placed over the quadriceps muscle.
  Other Names: -Bandages; -Tape; -Taping; -Kinesio Tex; -Kinesio Tape; -Kinesiotape
  Arms: Kinesio Taping; Kinesio Taping Placebo

SUMMARY:
Forty-eight female patients will be randomized into three groups to receive the Kinesio taping, placebo Kinesio taping and control group. The group Kinesio taping receive the correct application of the method described. The placebo group will receive a placement without tension. The control group did not receive any form of intervention.

DETAILED DESCRIPTION:
The group Kinesio taping receive the correct application of the method described with tension of 40%. The placebo group will receive a placement without tension.

The control group did not receive any form of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Sedentary

Exclusion Criteria:

* Physically active,
* pain
* men
* musculoskeletal injury in the last six months.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Vertical Jump | 40 minutes
  The vertical jump will be evaluated by the Counter Movement Jump

SECONDARY OUTCOMES:
Flexibility | 40 minutes
  The flexibility will be evaluate by fleximeter

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Luz, MSc, Principal Investigator — Paulista University
Locations (1):
- Universidade Paulista, Jundiaí, São Paulo, Brazil